CLINICAL TRIAL: NCT06256705
Title: Multi-modal Characterisation of Gastroenteropancreatic Neuroendocrine Tumours (GEP-NETs) Treated With Targeted Radionuclide Therapy (TRT): Prospective Interventional Multicentre National Cohort
Acronym: OPERANDI-NET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230280
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor; Radiotherapy
Keywords: Targeted radionuclide therapy
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-MRI (Experimental): PET-MRI added in care pathway
  Interventions: Other: Simultaneous 68Ga-DOTATOC PET-MRI

INTERVENTIONS:
Other: Simultaneous 68Ga-DOTATOC PET-MRI — on month before first cycle of 177Lu-DOTATATE, after second cycle and one year after first cycle

SUMMARY:
Operandi project aims to address unmet clinical needs in the current management of GEP-NETs treated with PRRT by exploring new opportunities provided by imaging-based (AI algorithms) and data augmentation, simultaneous 68Ga-DOTATOC PET-MRI imaging, and novel approaches to increase patient selection and PRRT efficacy (genomic profiling, radiopotentiators, and new radionuclides). The study aim to identify predictive and early markers indicative of PRRT effectiveness based on a large prospective cohort of GEP-NET patients. This cohort will be used to uncover relevant predictive signatures within the morphological, functional, and molecular imaging data using novel imaging-based AI approaches with a new patient imaging pathway including simultaneous 68Ga-DOTATOC PET-MRI.

Considering this global objective, the objective of this clinical research protocol is to provide clinical, molecular and imaging data in a prospective standardized study, notably by performing systematic PET-MRI at baseline, at mid course of PRRT and 1 year after PRRT initiation, in patients with advanced GEP-NETs treated with PRRT.

DETAILED DESCRIPTION:
Gastroenteropancreatic neuroendocrine tumours (GEP-NETs) are considered rare neoplasms. Their incidence has been increasing over the last few decades, and due to generally prolonged survival of patients, the prevalence of GEP-NETs is higher than the combined prevalence of other more common gastrointestinal cancers, including oesophageal cancers, gastric adenocarcinomas, and pancreatic adenocarcinomas. Prognosis is related to several factors and especially to liver tumour involvement.

Peptide Receptor Radionuclide Therapy (PRRT) is a targeted radionuclide therapy that has been used in the treatment of patients with GEP-NETs for over two decades. The molecular target for PRRT in NETs is the somatostatin receptor (SSTR), mainly the subtype 2, which is highly expressed in most of these tumours. The 177lu-DOTATATE, a radiolabelled somatostatin analog, has reached a wide use due to a combination of high anti-tumour activity and a low level of toxicity. 177Lu-DOTATATE was granted marketing authorisation by the European Medicines Agency in 2017 and by the Food and Drug Administration in 2018 for the treatment of GEP-NETs. Due to its high efficacy, it has become one of the most relevant therapeutic option for patients with inoperable and/or metastatic GEP-NETs.

Response evaluation - PRRT exerts antitumor effects based on radio-biological (DNA damages) and immunological mechanisms. While highly promising, patient stratification and early identification of responders are currently insufficient due to the lack of reliable biomarkers, either non-invasive or invasive. Furthermore, prior therapy-induced DNA damages may lead to tumour resistance, therefore reducing PRRT efficacy. Hence, the absence of a personalized treatment strategy is an unmet need for patients with GEP-NETs. This may result in survival disadvantage for non-responders, who could benefit otherwise from early treatment change, with expected more favourable outcomes.

Simultaneous PET-MRI: OPERANDI project proposes an innovative and holistic approach via PET-MRI guided therapy with somatostatin analogues (68Ga-DOTATOC). Our hypothesis is that simultaneous 68Ga-DOTATOC PET-MRI imaging provides more robust non-invasive predictive biomarkers than classical approach. This requires technological development of PET-MRI, with most methodological challenges being attenuation correction, reducing the impact of organ motion due to respiration and cardiac motion, and minimizing truncation and susceptibility artefacts.

A PET/MRI scan is a two-in-one exam that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan. This new hybrid technology harnesses the strengths of PET and MRI to produce some of the most highly detailed images currently available. MRI scans use a strong (1.5 to 3T for clinical use) magnetic field to produce detailed morphologic images and some sequences provide functioning information (such as diffusion-weighted, dynamic contrast-enhanced, MR elastography sequence). PET scan use radiotracers according to the clinical indications to highlight metabolism or biological changes.

The most common radiotracer that has been used so far is fluorodeoxyglucose (FDG), which detects metabolically active malignant lesions. Gallium-68-labeled somatostatin analogues (including 68Ga DOTATOC) are differentiation markers in NETs and are a prerequisite for verifying sufficient SSTR2 expression and selecting patients for PRRT.

The OPERANDI project aims to address unmet clinical needs in the current management of GEP-NETs treated with PRRT by exploring new opportunities provided by imaging-based (AI algorithms) and data augmentation, simultaneous 68Ga-DOTATOC PET-MRI imaging, and novel approaches to increase patient selection and PRRT efficacy (genomic profiling, radiopotentiators, and new radionuclides). The study aim to identify predictive and early markers indicative of PRRT effectiveness based on a large prospective cohort of GEP-NET patients. This cohort will be used to uncover relevant predictive signatures within the morphological, functional, and molecular imaging data using novel imaging-based AI approaches with a new patient imaging pathway including simultaneous 68Ga-DOTATOC PET-MRI.

ELIGIBILITY:
Inclusion Criteria:

* According the MDT decision to refer to PRRT

  1. Histologically confirmed diagnosis of unresectable GEP-NETs whatever the grade or NETs of unknown primary but suspected of GEP origin
  2. Metastastic and progressive according RECIST 1.1 criteria
  3. At least 1 measurable site of disease per RECIST v1.1 using contrast-enhanced CT or magnetic resonance imaging
  4. SSTR+ disease, as evidenced by PET-DOTATOC performed within 4 months prior to inclusion (lesion uptake greater than liver physiological uptake)
  5. The majority of the lesions and all RECIST 1.1 selected target lesion have to be SSTR+.
* Karnofsky performance status scale ≥ 60
* Live expectancy >6 months
* Patients ≥ 18 years of age

Exclusion Criteria:

* Known pregnancy or breastfeeding women
* Known hypersensitivity to 177Lu, octreotate, DOTA, 68Ga, Edotreotide,
* Known hypersensitivity to lysine, arginine, or any excipient of the nephroprotective amino acid solution (AAS) given concomitantly to the 177Lu-DOTATATE infusion.
* Contraindication to MRI and technical impossibility of MRI
* Prior external beam radiation therapy (EBRT) of GEP-NET lesions or liver selective internal radiation therapy within 12 weeks before inclusion, if extensive
* Other systemic antitumor treatment (non-radioactive, excluding somatostatin analogues) not interrupted for at least 4 weeks
* Mixed Neuroendocrine-Non-endocrine Neoplasms (MiNEN)
* Neuroendocrine carcinoma
* Uncontrolled brain metastasis for at least 3 months
* NYHA 3 or 4 heart failure
* Inability to discontinue delayed-acting somatostatin analogues at least 28 days prior the PRRT or rapid-acting somatostatin analogues at least 24 hours prior the PRRT
* Non-adequate bone marrow, liver and renal function within 1 month prior the PRRT as assessed by the following laboratory tests:

  * Platelet count < 75,000/mm3
  * Haemoglobin ≤ 8,0 g/dL
  * Total bilirubin > 3 ULN
  * Neutrophils < 1000/mm3
  * Prothrombin time < 70% unless albumin > 30g/L
  * Albumin <30g/L unless prothrombin time > 70 %
  * Glomerular Filtration Rate (GFR) < 35 mL/min/1.73 m2
* Prior peptide receptor radionuclide therapy (PRRT)
* Other progressive cancer excluding in situ cervical cancer and basal or squamous cell skin cancer within the last 3 years
* Patient refusal to give written informed consent
* Subject deprived of freedom, subject under a legal protective measure
* No affiliation to a social security regimen or CMU
* Patient under State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2028-03-25 (Estimated); Study Completion 2029-09-25 (Estimated)

PRIMARY OUTCOMES:
Clinical response defined by the PFS as the time measured from the day of first administration of PRRT to first progression or death at 18 months, whichever occurs first | 18 months after PRRT

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Médecine nucléaire et Biophysique - Beaujon, Clichy
  - Pancréatologie et Oncologie Digestive - Beaujon, Clichy
  - Hépato-gastro-entérologie, cancérologie digestive et assistance nutritionnelle - CHU Nantes, Nantes
  - Médecine nucléaire - CHU Nantes, Nantes
  - Service de Médecine Nucléaire, Groupe Hospitalier Bichat-Claude Bernard, Paris